CLINICAL TRIAL: NCT04582266
Title: Pharmacokinetics and Safety of Remdesivir for Treatment of COVID-19 in Pregnant and Non-Pregnant Women in the United States
Brief Title: PK and Safety of Remdesivir for Treatment of COVID-19 in Pregnant and Non-Pregnant Women in the US
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: IMPAACT 2032; DAIDS Study ID 38746 (Other: DAIDS CRMS)
Record Dates: First submitted 2020-10-08; First posted 2020-10-09 (Actual); Results first posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: COVID-19, Pregnancy
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Arm 1: Pregnant women hospitalized and receiving RDV for treatment of COVID-19.
  Interventions: Drug: Remdesivir
- Arm 2: Non-pregnant women of childbearing potential hospitalized and receiving RDV for treatment of COVID-19.
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Remdesivir — RDV was not provided as part of the study. Participants were administered RDV intravenously once daily for up to 10 days per clinical care.

SUMMARY:
IMPAACT 2032 was a Phase IV prospective, open label, non-randomized opportunistic study. The objectives of this study were to describe the pharmacokinetic (PK) properties and safety of remdesivir (RDV) administered intravenously as part of clinical care among hospitalized pregnant and non-pregnant women of childbearing potential with coronavirus disease of 2019 (COVID-19). RDV was provided and managed by the participant's treating physician and was not provided as part of this study.

DETAILED DESCRIPTION:
IMPAACT 2032 was a Phase IV prospective, open label, non-randomized opportunistic study to evaluate the PK and safety of RDV when administered to pregnant and non-pregnant women of childbearing potential for treatment of COVID-19. Participants were pregnant and non-pregnant women hospitalized for COVID-19 who received daily RDV infusions, typically for 5 days but in some cases for up to 10 days, as part of their clinical care. RDV was provided and managed by the participants' treating physician and was not provided as a part of this study.

This study was comprised of two population-based arms: Arm 1 included pregnant women of any gestational age (GA) and Arm 2 included non-pregnant women of childbearing potential, who were between 18 and 45 years of age. The target sample size was 20 PK-evaluable participants per arm. Study sites were located in the United States.

Study procedures for this study were limited to data collection and blood specimens for PK. Except for PK sampling, study procedures were largely done via medical chart abstraction or remote contact/telemedicine visit. Collection of clinical and laboratory data started at 48 hours before the first infusion and continued through 4 weeks after the last infusion. In addition, data were collected at the time of delivery for participants in Arm 1, and limited data were also collected from the birth and newborn exam records of their infants. All participants were followed for safety through 4 weeks after the last infusion; Arm 1 participants who were still pregnant at that time had an additional follow-up at the time of delivery. If there was a gap in time between 4 weeks after the last infusion and delivery, no data were collected during that interval.

No formal statistical comparisons were made between Arm 1 and Arm 2 for primary and secondary objectives. Therefore, all analyses for primary and secondary outcome measures represent single arm evaluations.

ELIGIBILITY:
Inclusion Criteria: Arm 1 (Pregnant Women)

* Of legal age or otherwise able to provide independent informed consent or is unable to provide informed consent (e.g., impaired capacity) and a Legally Authorized Representative (LAR) is willing and able to provide written informed consent on behalf of the participant
* At study entry, viable intra-uterine pregnancy of any gestational age, based on medical records.
* At study entry, hospitalized AND has confirmed or suspected COVID-19, based on medical records.
* At study entry, receiving or expected to receive RDV for COVID-19 clinical care, as prescribed by the clinical care provider and documented in medical records.

Inclusion Criteria - Arm 2 (Non-Pregnant Women)

* Of legal age or otherwise able to provide independent informed consent or is unable to provide informed consent (e.g., impaired capacity) and a Legally Authorized Representative (LAR) is willing and able to provide written informed consent on behalf of the participant
* At study entry, between 18 and 45 years of age, based on medical records and participant report.
* Assigned female at birth and at study entry not taking cross-sex hormone therapy.
* At study entry, not suspected to be pregnant, based on participant report and/or investigator or designee determination.
* At study entry, hospitalized AND has confirmed or suspected COVID-19, based on medical records.
* At study entry, receiving or expected to receive RDV for COVID-19 clinical care, as prescribed by the clinical care provider and documented in medical records.

Exclusion Criteria:

* At study entry, has started or received the 4th RDV infusion.
* At study entry, evidence of post-menopausal status (medical or surgical), based on medical records and/or participant report.
* At study entry, any contraindications to RDV treatment for COVID-19, based on investigator or designee determination.
* Received or administered any disallowed medications within 48 hours prior to study entry.
* At study entry, has any other condition, that, in the opinion of the site investigator or designee, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving study objectives.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study was conducted among hospitalized pregnant and non-pregnant women receiving RDV for treatment of COVID-19 as part of their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Mirochnick, MD, Study Chair — Department of Pediatrics, Boston University Chobanian and Avedisian School of Medicine; Diana Clarke, PharmD, Study Chair — Pediatric Infectious Diseases, Boston Medical Center; Brookie Best, PharmD, MAS, Study Chair — University of California, San Diego
Locations (10):
- United States (10):
  - David Geffen School of Medicine at UCLA (Site #: 5112), Los Angeles, California
  - Childrens Hospital (U. Colorado, Denver) NICHD CRS (Site #: 5052), Denver, Colorado
  - Pediatric Perinatal HIV Clinical Trials Unit (Site #: 5127), Miami, Florida
  - Emory University School of Medicine (Site #: 5030), Atlanta, Georgia
  - Rush University Cook County Hospital NICHD CRS (Site #: 5083), Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS (Site #: 4001), Chicago, Illinois
  - Johns Hopkins University NICHD CRS (Site #: 5092), Baltimore, Maryland
  - Stony Brook University Medical Center (Site #: 5040), Stony Brook, New York
  - Bronx-Lebanon Hospital Center (Site #: 5114), The Bronx, New York
  - Texas Children's Hospital (Site #: 5128), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/resources/study-proposals.htm. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.
URL: https://www.impaactnetwork.org/

REFERENCES:
- [Derived] Brooks KM, Baltrusaitis K, Clarke DF, Nachman S, Jao J, Purswani MU, Agwu A, Beneri C, Deville JG, Powis KM, Stek AM, Eke AC, Shapiro DE, Capparelli E, Greene E, George K, Yin DE, Jean-Philippe P, Chakhtoura N, Bone F, Bacon K, Johnston B, Reding C, Kersey K, Humeniuk R, Best BM, Mirochnick M, Momper JD; IMPAACT 2032 Study Team. Pharmacokinetics and Safety of Remdesivir in Pregnant and Nonpregnant Women With COVID-19: Results From IMPAACT 2032. J Infect Dis. 2024 Oct 16;230(4):878-888. doi: 10.1093/infdis/jiae298. PMID 38839047
- See also: DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, dated July 2017 — http://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment methods for this study relied on identification of pregnant and non-pregnant women hospitalized for coronavirus disease of 2019 (COVID-19) in a facility that is affiliated with an IMPAACT clinical research site and who recently initiated treatment with remdesivir (RDV) or who may require treatment with RDV. Enrollment occurred between March 31, 2021 and December 29, 2021 across ten sites in the United States.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 26 | 28
Received RDV | 25 | 28
Completed | 17 | 23
Not Completed | 9 | 5
Not completed — Lost to Follow-up | 7 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Logistical and Personnel Constraints at Time of Infusion | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population included all women who received any amount of RDV.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 25 | 28 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.2 (6.4) | 35.3 (7.4) | 33.8 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 28 | 53
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 6 | 18
  Not Hispanic or Latino | 12 | 17 | 29
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 16 | 22
  White | 10 | 6 | 16
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 25 | 28 | 53

OUTCOME MEASURES:

1. Primary Outcome: PK Outcome: Geometric Mean Area Under the Plasma Concentration-time Curve (AUC) of Remdesivir (RDV) in Arm 1
Description: AUC calculated using non-compartmental methods with linear up-log down trapezoidal rule (Phoenix WinNonlin v 8.3, Certara®). Intensive PK sampling occurred once, on the day of the 3rd, 4th, or 5th infusion.
Time Frame: At 3rd, 4th, or 5th infusion. Collection timepoints included: pre-dose, end of infusion (EOI), EOI + 0.75 hours, EOI + 1.5 hours, EOI + 3 hours, EOI + 5 hours, EOI + 7 hours, EOI + 23 hours.
Population: Arm 1 women who met the following minimum sampling requirements: (1) at least 3 out of 4 of the end of infusion (EOI) through 3 hours post-end-of-infusion (post-EOI) intensive PK samples AND (2) either the 5 hours post-EOI or the 7 hours post-EOI intensive PK sample AND (3) either the pre-dose or 23-hour post-EOI intensive PK sample, had at least two drug concentrations greater than the lower limit of quantification, and had an available RDV AUC measurement.
Measure: Geometric Mean (90% Confidence Interval); unit: h*ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 18
h*ng/mL | 1246.57 [915.71 to 1696.99]

2. Primary Outcome: PK Outcome: Geometric Mean Half-life (t1/2) of Remdesivir (RDV) in Arm 1
Description: t1/2 calculated using non-compartmental methods with linear up-log down trapezoidal rule (Phoenix WinNonlin v 8.3, Certara®). Intensive PK sampling occurred once, on the day of the 3rd, 4th, or 5th infusion.
Time Frame: as for outcome 1
Population: Arm 1 women who met the following minimum sampling requirements: (1) at least 3 out of 4 of the end of infusion (EOI) through 3 hours post-end-of-infusion (post-EOI) intensive PK samples AND (2) either the 5 hours post-EOI or the 7 hours post-EOI intensive PK sample AND (3) either the pre-dose or 23-hour post-EOI intensive PK sample, had at least two drug concentrations greater than the lower limit of quantification, and had an available RDV t1/2 measurement.
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Arm/Group | Arm 1
Number analyzed (Participants) | 17
hours | 1.01 [0.87 to 1.17]

3. Primary Outcome: PK Outcome: Geometric Mean Trough Concentration (Ctrough) of GS-441524 in Arm 1
Description: GS-441524 is a metabolite of remdesivir (RDV). Ctrough calculated using non-compartmental methods with linear up-log down trapezoidal rule (Phoenix WinNonlin v 8.3, Certara®). Intensive PK sampling occurred once, on the day of the 3rd, 4th, or 5th infusion.
Time Frame: as for outcome 1
Population: Arm 1 women who met the following minimum sampling requirements: (1) at least 3 out of 4 of the end of infusion (EOI) through 3 hours post-end-of-infusion (post-EOI) intensive PK samples AND (2) either the 5 hours post-EOI or the 7 hours post-EOI intensive PK sample AND (3) either the pre-dose or 23-hour post-EOI intensive PK sample, had at least two drug concentrations greater than the lower limit of quantification, and had an available GS-441524 Ctrough measurement.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Arm 1
Number analyzed (Participants) | 20
ng/mL | 51.6 [44.7 to 59.6]

4. Primary Outcome: Safety Outcome: Proportion of Participants With Maternal Renal Adverse Event (AE) of Any Grade in Arm 1
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one maternal renal AE through 7 days post last infusion, bounded by an exact 95% confidence interval (CI). Renal AEs were defined using the MedDRA system organ class term "Renal and urinary disorders" and high level grouping term "Renal and urinary tract investigations and urinalyses". The number of RDV infusions varied by participant.
Time Frame: First infusion through 7 Days post-last infusion
Population: Arm 1 women who receive any amount of RDV and had follow-up through 7 days post-last infusion or a renal adverse event of any grade.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 23
proportion of participants | 0 [0 to 0.15]

5. Primary Outcome: Safety Outcome: Proportion of Participants With Maternal Hepatic Adverse Event (AE) of Any Grade in Arm 1
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one maternal hepatic AE through 7 days post last infusion, bounded by an exact 95% confidence interval (CI). Hepatic AEs were defined using the MedDRA system organ class term "Hepatobiliary disorders" and high level grouping term "Hepatobiliary investigations". The number of RDV infusions varied by participant.
Time Frame: First infusion through 7 Days post-last infusion
Population: Arm 1 women who receive any amount of RDV and had follow-up through 7 days post-last infusion or a hepatic adverse event of any grade.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 23
proportion of participants | 0.04 [0.00 to 0.22]

6. Primary Outcome: Safety Outcome: Proportion of Participants With Maternal Hematologic Adverse Event (AE) of Any Grade in Arm 1
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one maternal hematologic AE through 7 days post last infusion, bounded by an exact 95% confidence interval (CI). Hematologic AEs were defined using the MedDRA system organ class term "Blood and lymphatic system disorders" and high level grouping term "Haematology investigations (incl blood groups)". The number of RDV infusions varied by participant.
Time Frame: First infusion through 7 Days post-last infusion
Population: Arm 1 women who receive any amount of RDV and had follow-up through 7 days post-last infusion or a hematologic adverse event of any grade.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 23
proportion of participants | 0.30 [0.13 to 0.53]

7. Primary Outcome: Safety Outcome: Proportion of Participants With Maternal Grade 3 or Higher Adverse Event (AE) in Arm 1
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one maternal grade 3 or higher adverse event through 4 weeks post last infusion and delivery, bounded by an exact 95% confidence interval (CI). The number of RDV infusions varied by participant.
Time Frame: First infusion through 4 Weeks post-last infusion and Delivery
Population: Arm 1 women who receive any amount of RDV and had follow-up through 4 weeks post-last infusion and delivery or at least one maternal grade 3 or higher adverse event.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 22
proportion of participants | 0.68 [0.45 to 0.86]

8. Primary Outcome: Safety Outcome: Proportion of Participants With Serious Adverse Event (AE) in Arm 1
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one maternal serious AE through 4 weeks post last infusion and delivery, bounded by an exact 95% confidence interval (CI). The number of RDV infusions varied by participant.
Time Frame: First infusion through 4 Weeks post-last infusion and Delivery
Population: Arm 1 women who receive any amount of RDV and had follow-up through 4 weeks post-last infusion and delivery or at least one maternal serious adverse event.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 18
proportion of participants | 0.33 [0.13 to 0.59]

9. Primary Outcome: Safety Outcome: Proportion of Participants With Maternal Grade 3 or Higher Adverse Event (AE) Assessed as Related to Remdesivir (RDV) by the Clinical Management Committee (CMC) in Arm 1
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one maternal grade 3 or higher AE assessed as related to RDV by the CMC through 4 weeks post last infusion and delivery, bounded by an exact 95% confidence interval (CI). The number of RDV infusions varied by participant.
Time Frame: First infusion through 4 Weeks post-last infusion and Delivery
Population: Arm 1 women who receive any amount of RDV and had follow-up through 4 weeks post-last infusion and delivery or at least one maternal grade 3 or higher adverse event assessed as related to RDV by the CMC.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 16
proportion of participants | 0.00 [0.00 to 0.21]

10. Primary Outcome: Safety Outcome: Proportion of Participants With Pregnancy Loss in Arm 1
Description: We present the proportion of participants who had a pregnancy loss at delivery, bounded by an exact 95% confidence interval (CI).
Time Frame: Delivery
Population: Arm 1 women who receive any amount of RDV and had a delivery visit.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 17
proportion of participants | 0.06 [0.00 to 0.29]

11. Primary Outcome: Safety Outcome: Proportion of Participants With Congenital Anomalies in Arm 1
Description: We present the proportion of participants who had a live infant born with congenital anomalies at delivery, bounded by an exact 95% confidence interval (CI).
Time Frame: Delivery
Population: Arm 1 women who receive any amount of RDV, had a delivery visit, and had a live-born infant.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 16
proportion of participants | 0.00 [0.00 to 0.21]

12. Primary Outcome: Safety Outcome: Proportion of Participants With Preterm Birth, Defined as < 37 Weeks in Arm 1
Description: We present the proportion of participants who had a live preterm birth defined as < 37 weeks, bounded by an exact 95% confidence interval (CI).
Time Frame: Delivery
Population: Arm 1 women who receive any amount of RDV, had a delivery visit, and had a live-born infant.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 16
proportion of participants | 0.25 [0.07 to 0.52]

13. Primary Outcome: Safety Outcome: Proportion of Participants With Preterm Birth, Defined as < 34 Weeks in Arm 1
Description: We present the proportion of participants who had a live preterm birth defined as < 34 weeks, bounded by an exact 95% confidence interval (CI).
Time Frame: Delivery
Population: Arm 1 women who receive any amount of RDV, had a delivery visit, and had a live-born infant.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 16
proportion of participants | 0.00 [0.00 to 0.21]

14. Primary Outcome: Safety Outcome: Proportion of Participants With Small for Gestational Age, Defined as < 10th Percentile in Arm 1
Description: We present the proportion of participants who a live born infant who was small for gestational age defined as < 10th percentile, bounded by an exact 95% confidence interval (CI).
Time Frame: Delivery
Population: Arm 1 women who receive any amount of RDV, had a delivery visit, and had a live-born infant.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 1
Number analyzed (Participants) | 16
proportion of participants | 0.13 [0.02 to 0.38]

15. Primary Outcome: Safety Outcome: Mean Newborn Birth Weight in Arm 1
Description: We present the newborn mean weight among the participants who had live born infant, bounded by a 95% confidence interval (CI) calculated using the t distribution.
Time Frame: Delivery
Population: Infants born to Arm 1 women, who received any amount of RDV and had a delivery visit, and had available weight measurement.
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | Arm 1
Number analyzed (Participants) | 16
kg | 3.039 [2.766 to 3.313]

16. Primary Outcome: Safety Outcome: Mean Newborn Length in Arm 1
Description: We present the newborn mean length among the participants who had a live born infant, bounded by a 95% confidence interval (CI) calculated using the t distribution.
Time Frame: Delivery
Population: Infants born to Arm 1 women, who received any amount of RDV and had a delivery visit, and had available length measurement.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Arm 1
Number analyzed (Participants) | 8
cm | 44.1 [37.1 to 51.1]

17. Primary Outcome: Safety Outcome: Mean Newborn Head Circumference in Arm 1
Description: We present the newborn mean head circumference among the participants who had a live born infant, bounded by a 95% confidence interval (CI) calculated using the t distribution.
Time Frame: Delivery
Population: Infants born to Arm 1 women, who received any amount of RDV and had a delivery visit, and had available head circumference measurement.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Arm 1
Number analyzed (Participants) | 8
cm | 29.9 [25.3 to 34.5]

18. Secondary Outcome: PK Outcome: Geometric Mean Area Under the Plasma Concentration-time Curve (AUC) of Remdesivir (RDV) in Arm 2
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Arm 2 women who met the following minimum sampling requirements: (1) at least 3 out of 4 of the end of infusion (EOI) through 3 hours post-end-of-infusion (post-EOI) intensive PK samples AND (2) either the 5 hours post-EOI or the 7 hours post-EOI intensive PK sample AND (3) either the pre-dose or 23-hour post-EOI intensive PK sample, had at least two drug concentrations greater than the lower limit of quantification, and had an available RDV AUC measurement.
Measure: Geometric Mean (90% Confidence Interval); unit: h*ng/mL
Arm/Group | Arm 2
Number analyzed (Participants) | 17
h*ng/mL | 1302.75 [1069.70 to 1586.58]

19. Secondary Outcome: PK Outcome: Geometric Mean Half-life (t1/2) of Remdesivir (RDV) in Arm 2
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Arm 2 women who met the following minimum sampling requirements: (1) at least 3 out of 4 of the end of infusion (EOI) through 3 hours post-end-of-infusion (post-EOI) intensive PK samples AND (2) either the 5 hours post-EOI or the 7 hours post-EOI intensive PK sample AND (3) either the pre-dose or 23-hour post-EOI intensive PK sample, had at least two drug concentrations greater than the lower limit of quantification, and had an available RDV t1/2 measurement.
Measure: Geometric Mean (90% Confidence Interval); unit: hours
Arm/Group | Arm 2
Number analyzed (Participants) | 16
hours | 1.09 [0.94 to 1.27]

20. Secondary Outcome: PK Outcome: Geometric Mean Trough Concentration (Ctrough) of GS-441524 in Arm 2
Description: as for outcome 3
Time Frame: as for outcome 1
Population: Arm 2 women who met the following minimum sampling requirements: (1) at least 3 out of 4 of the end of infusion (EOI) through 3 hours post-end-of-infusion (post-EOI) intensive PK samples AND (2) either the 5 hours post-EOI or the 7 hours post-EOI intensive PK sample AND (3) either the pre-dose or 23-hour post-EOI intensive PK sample, had at least two drug concentrations greater than the lower limit of quantification, and had an available GS-441524 Ctrough measurement.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Arm 2
Number analyzed (Participants) | 21
ng/mL | 57.1 [48.7 to 66.9]

21. Secondary Outcome: Safety Outcome: Proportion of Participants With Renal Adverse Event (AE) of Any Grade in Arm 2
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one renal AE through 7 days post last infusion, bounded by an exact 95% confidence interval (CI). Renal AEs were defined using the MedDRA system organ class term "Renal and urinary disorders" and high level grouping term "Renal and urinary tract investigations and urinalyses". The number of RDV infusions varied by participant.
Time Frame: First infusion through 7 Days post-last infusion
Population: Arm 2 women who receive any amount of RDV and had follow-up through 7 days post-last infusion or a renal adverse event of any grade.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 2
Number analyzed (Participants) | 23
proportion of participants | 0.04 [0.00 to 0.22]

22. Secondary Outcome: Safety Outcome: Proportion of Participants With Hepatic Adverse Event (AE) of Any Grade in Arm 2
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one hepatic AE through 7 days post last infusion, bounded by an exact 95% confidence interval (CI). Hepatic AEs were defined using the MedDRA system organ class term "Hepatobiliary disorders" and high level grouping term "Hepatobiliary investigations". The number of RDV infusions varied by participant.
Time Frame: First infusion through 7 Days post-last infusion
Population: Arm 2 women who receive any amount of RDV and had follow-up through 7 days post-last infusion or a hepatic adverse event of any grade.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 2
Number analyzed (Participants) | 24
proportion of participants | 0.04 [0.00 to 0.21]

23. Secondary Outcome: Safety Outcome: Proportion of Participants With Hematologic Adverse Event (AE) of Any Grade in Arm 2
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one hematologic AE through 7 days post last infusion, bounded by an exact 95% confidence interval (CI). Hematologic AEs were defined using the MedDRA system organ class term "Blood and lymphatic system disorders" and high level grouping term "Haematology investigations (incl blood groups)". The number of RDV infusions varied by participant.
Time Frame: First infusion through 7 Days post-last infusion
Population: Arm 2 women who receive any amount of RDV and had follow-up through 7 days post-last infusion or a hematologic adverse event of any grade.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 2
Number analyzed (Participants) | 23
proportion of participants | 0.26 [0.10 to 0.48]

24. Secondary Outcome: Safety Outcome: Proportion of Participants With Grade 3 or Higher Adverse Event (AE) in Arm 2
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE through 4 weeks post last infusion, bounded by an exact 95% confidence interval (CI).
Time Frame: First infusion through 4 Weeks post-last infusion
Population: Arm 2 women who receive any amount of RDV and had follow-up through 4 weeks post-last infusion or at least one grade 3 or higher adverse event.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 2
Number analyzed (Participants) | 24
proportion of participants | 0.54 [0.33 to 0.74]

25. Secondary Outcome: Safety Outcome: Proportion of Participants With Serious Adverse Event (AE) in Arm 2
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. We present the proportion of participants with at least one serious AE through 4 weeks post last infusion, bounded by an exact 95% confidence interval (CI). The number of RDV infusions varied by participant.
Time Frame: First infusion through 4 Weeks post-last infusion
Population: Arm 2 women who receive any amount of RDV and had follow-up through 4 weeks post-last infusion or at least one serious adverse event.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 2
Number analyzed (Participants) | 23
proportion of participants | 0.17 [0.05 to 0.39]

26. Secondary Outcome: Safety Outcome: Proportion of Participants With Grade 3 or Higher Adverse Event (AE) Assessed as Related to Remdesivir (RDV) by the Clinical Management Committee (CMC) in Arm 2
Description: Graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. The DAIDS grading table provides an AE severity grading scale ranging from grades 1 to 5 with descriptions for each AE based on the following general guidelines: grade 1 indicates a mild event, grade 2 indicates a moderate event, grade 3 indicates a severe event, grade 4 indicates a potentially life-threatening event, and grade 5 indicates death. We present the proportion of participants with at least one grade 3 or higher AE as related to RDV by the CMC through 4 weeks post last infusion, bounded by an exact 95% confidence interval (CI). The number of RDV infusions varied by participant.
Time Frame: First infusion through 4 Weeks post-last infusion
Population: Arm 2 women who receive any amount of RDV and had follow-up through 4 weeks post-last infusion or at least one grade 3 or higher adverse event assess as related to RDV by the CMC.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm 2
Number analyzed (Participants) | 23
proportion of participants | 0.04 [0.00 to 0.22]

27. Other Pre Specified Outcome: PK Outcome: Ratio of Cord Blood/Maternal Plasma Remdisivir (RDV) Concentrations
Description: Ratio of cord blood/maternal plasma is calculated for women in Arm 1 who received RDV within 5 days of delivery only.
Time Frame: Delivery
Population: No cord blood was collected.
Arm/Group | Arm 1
Number analyzed (Participants) | 0

28. Other Pre Specified Outcome: PK Outcome: Ratio of Cord Blood/Maternal Plasma GS-441524 Concentrations
Description: GS-441524 is a metabolite of remdesivir (RDV). Ratio of cord blood/maternal plasma is calculated for women in Arm 1 who received RDV within 5 days of delivery only.
Time Frame: Delivery
Population: No cord blood was collected.
Arm/Group | Arm 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Enrolled women in Arm 1 were followed for 4 weeks after the last RDV infusion and at delivery. Enrolled women in Arm 2 were followed for 4 weeks after the last RDV infusion.
Description: The definition of adverse event provided in Version 2.0 of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual) was used in this study. This definition was applied to all participants at the time of the first infusion until four weeks after the last infusion and during the Delivery period for Arm 1 participants, if it occurred after Safety Follow-up period. Any medical conditions that occurred prior to the first infusion were considered pre-existing conditions.
Arm/Group | Arm 1 | Arm 2
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/28
Serious Adverse Events (participants affected / at risk) | 7/25 | 4/28
Other Adverse Events (participants affected / at risk) | 15/25 | 15/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=25) | Arm 2 (N=28)
Foetal heart rate deceleration abnormality (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Superimposed pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (N=25) | Arm 2 (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2
Bradycardia (Cardiac disorders) | 0 | 1
Left ventricular dilatation (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Infusion site oedema (General disorders) | 1 | 0
Infusion site pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 3 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 2
Blood pressure increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 4 | 1
International normalised ratio increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 4 | 1
Oxygen saturation decreased (Investigations) | 2 | 0
Prothrombin time prolonged (Investigations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
High risk pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Large for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Premature delivery (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 3 | 0
Jugular vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Because the study population might not include women who started RDV and discontinued it before the fourth infusion, this study may not identify PK, safety, or tolerance issues that occur after drug initiation and estimates of the frequency of adverse outcomes might be optimistic. Due to the way the data was collected, some AEs may not have been detected following hospital discharge.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT04582266/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2022-04-11): https://cdn.clinicaltrials.gov/large-docs/66/NCT04582266/SAP_001.pdf